CLINICAL TRIAL: NCT01120964
Title: Phase IB Double Blind, Randomized, Placebo Controlled Clinical Trial to Determine the Pharmacokinetics and Safety of a Revised Protocol of Intravenous L-Citrulline (Citrupress®) Versus Placebo in Children Undergoing Cardiopulmonary Bypass
Brief Title: Intravenous L-Citrulline to Treat Children Undergoing Heart Bypass Surgery : Revised Protocol
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Asklepion Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CIT-002-01
Record Dates: First submitted 2010-05-06; First posted 2010-05-11 (Estimated); Results first posted 2022-06-21 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Atrial Septal Defect; Ventricular Septal Defect; Atrioventricular Septal Defect
MeSH Terms: conditions — Heart Septal Defects, Atrial; Heart Septal Defects, Ventricular; Atrioventricular Septal Defect

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous L-Citrulline (Experimental): IV bolus of 150 mg/kg L-citrulline at the initiation of bypass, followed by L-citrulline (200 μmol/L) addition to the filtration or hemoconcentration replacement fluid used during bypass. Plus L-citrulline (20 mg/kg) bolus 30 minutes after decannulation from bypass, immediately followed by 9 mg/kg/h continuous L-citrulline infusion for 48 hours.
  Interventions: Drug: Intravenous L-Citrulline
- Placebo of Intravenous L-Citrulline (Placebo Comparator): Placebo administered according to the same schedule as L-citrulline
  Interventions: Drug: Placebo of Intravenous L-Citrulline

INTERVENTIONS:
Drug: Intravenous L-Citrulline
  Arms: Intravenous L-Citrulline
Drug: Placebo of Intravenous L-Citrulline — Placebo of intravenous L-Citrulline given at the same prescribed times as L-Citrullne Drug
  Arms: Placebo of Intravenous L-Citrulline

SUMMARY:
This clinical trial will determine the safety and effectiveness of intravenous L-citrulline in children undergoing cardiopulmonary bypass during heart surgery. Participants will be randomly assigned to either L-citrulline or a placebo (a substance that has no medicine in it).

Citrulline is a protein building block in the body that can convert into another substance, nitric oxide (NO), which controls blood pressure in the lungs. Increased blood pressure in the lungs can be an important surgical problem; it may also lead to problems following surgery, such as severe high blood pressure in the lungs (pulmonary hypertension), increased time spent on a breathing machine, and a longer stay in the intensive care unit (ICU). The hypothesis of this study is that perioperative supplementation with intravenous citrulline will increase plasma citrulline, arginine and NO metabolites and prevent elevations in the postoperative PVT leading to a decrease in the duration of postoperative invasive mechanical ventilation.

The objective of this study is to determine in a randomized placebo controlled phase IB multicenter clinical trial if a revised protocol of intravenous L-citrulline delivery given perioperatively achieves a plasma citrulline level of > 100 umol/L in children undergoing surgical repair of an atrial septal defect,ventricular septal defect or an atrioventricular septal defect.

DETAILED DESCRIPTION:
Increased pulmonary vascular tone (PVT) can complicate the postoperative course of the following five surgical procedures for congenital heart defects: 1) unrestrictive ventricular septal defect (VSD) repair; 2) atrioventricular septal (AVSD) repair; 3) arterial switch procedure for transposition of the great arteries (TGA); 4) bidirectional Glenn shunt procedure; and 5) Fontan procedure for single ventricle lesions. PVT is partially controlled by NO. Arginine, the precursor to NO, is a product of the urea cycle. Preliminary data have been presented regarding 169 infants and children who have undergone one of six previous surgical procedures. It was found that urea cycle function and plasma arginine levels were significantly decreased in all participants. Furthermore, participants with increased PVT had significantly lower arginine levels compared to participants with normal PVT. Finally, a genetic single nucleotide polymorphism (SNP) in the rate limiting urea cycle enzyme (carbamyl phosphate synthetase I [CPSl T1405N]) appeared to affect postoperative plasma arginine levels and PVT. It is hypothesized that perioperative enhancement of urea cycle function with the key urea cycle intermediate (citrulline) will increase plasma arginine and NO metabolites and prevent elevations in PVT.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent signed by the subject's legal representative
2. Subjects < 6 years old
3. Subjects undergoing cardiopulmonary bypass for repair of an atrial septal defect, a ventricular septal defect or an atrioventricular septal defect

Exclusion Criteria:

1. Pulmonary artery or vein abnormalities being addressed surgically
2. Preoperative requirement for invasive mechanical ventilation or intravenous inotrope support
3. Any condition which, in the opinion of the investigator, might interfere with study objectives

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2010-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick E Barr, MD, Study Chair — Batson Children's Hospital, University of Mississippi Medical Center; Catherine Krawczeski, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Allan Doctor, MD, Principal Investigator — St. Louis Children's Medical Center
Locations (2):
- United States (2):
  - Washington University Children's Hospital, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravenous L-Citrulline: IV bolus of 150 mg/kg L-citrulline at the initiation of bypass, followed by L-citrulline (200 μmol/L) addition to the filtration or hemoconcentration replacement fluid used during bypass. Plus L-citrulline (20 mg/kg) bolus 30 minutes after decannulation from bypass, immediately followed by 9 mg/kg/h continuous L-citrulline infusion for 48 hours.
  Intravenous L-Citrulline
Period: Overall Study
Arm/Group | Intravenous L-Citrulline | Placebo of Intravenous L-Citrulline
Started | 11 | 11
Completed | 10 | 11
Not Completed | 1 | 0
Not completed — Did not receive full treatment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous L-Citrulline | Placebo of Intravenous L-Citrulline | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 11 | 22
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 28.5 (22.4) | 15.3 (17.1) | 21.9 (20.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 6 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 10 | 7 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: L-citrulline Plasma Levels
Description: Citrulline Blood Levels: 1. Baseline sample in OR prior to Cardiopulmonary Bypass prior to administration of first bolus of Citrulline or Placebo 2. Immediately after Bolus 1 administered in Operating Room. 3. 30 minutes after separation from Cardiopulmonary Bypass; immediately prior to administration of Bolus 2 and start of continuous infusion of Citrulline or Placebo. 4. Six hours after after start of infusion. 5. 12 hours after start of infusion. 6. 24 hours after start of infusion. 7. 48 hours after start of infusion; or whenever infusion is discontinued if prior to 48 hours.
Time Frame: Measured in seven blood sample time points from the beginning of surgery until end of IV Citrulline Infusion; at either 48 hours postoperatively or at extubation, whichever comes first.
Population: All randomized patients that received surgery, were treated with L-citrulline, and had at least 1 citrulline concentration measurement
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Intravenous L-Citrulline | Placebo of Intravenous L-Citrulline
Number analyzed (Participants) | 11 | 11
µmol/L
  Baseline | 200.9 (569.89) | 34.1 (7.5)
  Post Bolus 1 | 2405.9 (1517.4) | 29.5 (5.96)
  Pre Bolus 2 | 890.9 (1077.5) | 30.6 (10.46)
  Hour 6: number analyzed (Participants) | 10 | 11
  Hour 6 | 167.8 (117.67) | 24.1 (7.76)
  Hour 12: number analyzed (Participants) | 10 | 9
  Hour 12 | 127.1 (16.18) | 19.9 (7.01)
  Hour 24 | 125.3 (38.74) | 12.9 (2.89)
  Hour 48: number analyzed (Participants) | 0 | 11
  Hour 48 |  | 12.3 (3.4)

2. Secondary Outcome: Postoperative Invasive Mechanical Ventilation (Mean and SD)
Description: Duration of postoperative invasive mechanical ventilation was derived as the time in hours from separation from cardiopulmonary bypass until endotracheal extubation. If a patient required reintubation within 24 hours after extubation, the reintubation time was added in the main analysis. In a second analysis, the reintubation time was not included.
Time Frame: Measured in hours from the end of surgery until extubation, or Day 30, whichever occurs first
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Intravenous L-Citrulline | Placebo of Intravenous L-Citrulline
Number analyzed (Participants) | 11 | 11
Hours
  Re-intubation time included | 5.1 (8.15) | 37.1 (65.41)
  Re-intubation time excluded | 5.1 (8.15) | 24.7 (26.83)
Statistical Analysis 1: Comparison: Intravenous L-Citrulline vs Placebo of Intravenous L-Citrulline; Total duration of postoperative invasive mechanical ventilation was analyzed by treatment group using summary statistics, and was compared between citrulline and placebo groups using an ANOVA. Kaplan-Meier analyses were performed for: 1) zero durations censored, 2) zero durations uncensored, 3) patients with zero duration excluded. The same analyses were performed with re-intubation time removed; Test type: Other — Analyses presented herein are for re-intubation time included; p = 0.0222, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p<0.05; Mean Difference (Final Values) = 32.0, 95% CI 2-sided [-9.5 to 73.4]

3. Secondary Outcome: Postoperative Invasive Mechanical Ventilation (Median and Range)
Description: as for outcome 2
Time Frame: Measured in hours from the end of surgery until extubation or Day 30, whichever occurred first
Measure: Median (Full Range); unit: Hours
Arm/Group | Intravenous L-Citrulline | Placebo of Intravenous L-Citrulline
Number analyzed (Participants) | 11 | 11
Hours
  Re-intubation time included | 0.0 [0.0 to 22.5] | 21.7 [0.0 to 229.3]
  Re-intubation time excluded | 0.0 [0.0 to 22.5] | 21.7 [0.0 to 92.3]
Statistical Analysis 1: Comparison: Intravenous L-Citrulline vs Placebo of Intravenous L-Citrulline; Analyses presented herein are for re-intubation time included; Test type: Other; p = 0.0222, t-test, 2 sided — Re-intubation time included. Threshold for significance was p<0.05; Mean Difference (Final Values) = 32.0, 95% CI 2-sided [-9.5 to 73.4]

4. Secondary Outcome: Total Duration of Respiratory Support
Description: Analysis included any invasive and non-invasive respiratory support required during the study period
Time Frame: Baseline to discharge or Day 30, whichever occurs first
Population: All randomized patients that received surgery
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Intravenous L-Citrulline | Placebo of Intravenous L-Citrulline
Number analyzed (Participants) | 11 | 11
Hours | 31.2 (28.27) | 81.9 (66.23)
Statistical Analysis 1: Comparison: Intravenous L-Citrulline vs Placebo of Intravenous L-Citrulline; Test type: Other; p = 0.0418, Wilcoxon (Mann-Whitney) — The threshold for significance was P<0.05; Mean Difference (Final Values) = 50.7, 95% CI 2-sided [5.4 to 96.0]

5. Secondary Outcome: Postoperative Intravenous Inotrope Duration
Description: The length of time on IV inotropes was documented from the time of first use after surgery until completion of the study medication at Hour 48 (i.e., duration of inotrope use was maximally 48 hours). Patients still receiving inotropes at Hour 48 were censored.
Time Frame: Measured at 48 hours
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Intravenous L-Citrulline | Placebo of Intravenous L-Citrulline
Number analyzed (Participants) | 11 | 11
Hours | 13.4 (14.78) | 26.1 (23.0)
Statistical Analysis 1: Comparison: Intravenous L-Citrulline vs Placebo of Intravenous L-Citrulline; Test type: Other; p = 0.0727, Wilcoxon (Mann-Whitney) — The threshold for significance was p<0.05; Mean Difference (Final Values) = 12.7, 95% CI 2-sided [-2.6 to 28.1]

6. Secondary Outcome: Total Inotrope Score
Description: The inotrope dose was calculated each hour postoperatively from the time of PICU admission until the completion of study drug using the following scoring system:
  Dopamine (μg/kg/min) x 1 plus Dobutamine (μg/kg/min) x 1 plus Milrinone (μg/kg/min) x10 plus Epinephrine (Adrenaline) (μg/kg/min) x 100 plus Phenylephrine (μg/kg/min) x 100 plus Norepinephrine (Noradrenaline) (μg/kg/min) x 100
  = Total inotrope score
  An ANOVA was performed. Additionally a repeated measures analysis of variance was used to compare total inotrope score between placebo and citrulline.
Time Frame: PICU admission until Hour 48
Measure: Mean (Standard Deviation); unit: µg/kg/min
Arm/Group | Intravenous L-Citrulline | Placebo of Intravenous L-Citrulline
Number analyzed (Participants) | 11 | 11
µg/kg/min | 602.7 (727.86) | 1162.6 (951.31)
Statistical Analysis 1: Comparison: Intravenous L-Citrulline vs Placebo of Intravenous L-Citrulline; Test type: Other; p = 0.1271, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 559.8, 95% CI 2-sided [-193.5 to 1313.2]

7. Secondary Outcome: Time on Vasoactive Medications
Description: The total number of hours on vasoactive medications, including nitroglycerin, nitroprusside and vasopressin, was calculated from the end of surgery until the discontinuation of vasoactive medications or end of study medication (Hour 48), whichever occurred first
Time Frame: Hour 0 to Hour 48
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Intravenous L-Citrulline | Placebo of Intravenous L-Citrulline
Number analyzed (Participants) | 11 | 11
Hours | 6.3 (7.18) | 9.8 (15.09)
Statistical Analysis 1: Comparison: Intravenous L-Citrulline vs Placebo of Intravenous L-Citrulline; Test type: Other; p = 0.9720, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 3.5, 95% CI 2-sided [-7.0 to 14.1]

8. Secondary Outcome: Total Vasoactive Score
Description: Vasoactive score is reflective of the pharmacological support required by the cardiovascular system and is a good predictor of mortality and morbidity in patients undergoing bypass surgery. A lower vasoactive score represents less pharmacological support and would indicate a lower risk for a poor clinical outcome. Therefore, any treatment effect would be indicated by a lower score in the citrulline group when compared to the placebo group.
  In this study, the score was calculated post-operatively from the time of separation from bypass until the completion of study drug. Vasoactive score was calculated using the following formula:
  Total Vasoactive Score = nitroglycerin dose + nitroprusside dose + vasopressin dose
  The minimum value is zero (i.e., no vasoactive drugs administered), but it is not possible to define a maximum as this is wholly dependent upon the dose of each vasoactive drug administered.
Time Frame: Hour 0 to Hour 48
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Intravenous L-Citrulline | Placebo of Intravenous L-Citrulline
Number analyzed (Participants) | 11 | 11
Score on a scale | 5.5 (10.62) | 10.6 (17.42)
Statistical Analysis 1: Comparison: Intravenous L-Citrulline vs Placebo of Intravenous L-Citrulline; Test type: Other; p = 0.8884, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 5.2, 95% CI 2-sided [-7.7 to 18.0]

9. Secondary Outcome: Length of ICU Stay
Description: Duration of ICU stay was analyzed once as the total number of postoperative hours spent in the ICU and once as the total number of postoperative hours that a patient required postoperative mechanical ventilator or continuous intravenous inotrope or vasodilator support. The latter combination of parameters represents another surrogate endpoint for ICU stay
Time Frame: Measured in hours from the end of surgery to discharge from ICU or Day 30, whichever occurred first
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Intravenous L-Citrulline | Placebo of Intravenous L-Citrulline
Number analyzed (Participants) | 11 | 11
Hours
  Duration of PICU stay | 35.94 (16.150) | 105.08 (187.762)
  Longest duration of mechanical ventilation, IV inotrope or vasodilator use (re-intubation included) | 14.5 (13.99) | 44.4 (63.62)
  Longest duration of mechanical ventilation, IV inotrope or vasodilator use (re-intubation excluded) | 14.5 (13.99) | 32.0 (26.26)
Statistical Analysis 1: Comparison: Intravenous L-Citrulline vs Placebo of Intravenous L-Citrulline; Test type: Other — Total number of postoperative hours spent in PICU; p = 0.1891, Wilcoxon (Mann-Whitney) — The threshold for significance was p<0.05; Mean Difference (Final Values) = 69.14, 95% CI 2-sided [-49.39 to 187.67]

10. Secondary Outcome: Composite Endpoint: Cessation of Positive Pressure Ventilation and of Inotrope Therapy
Description: The composite endpoint comprised the longer of the duration of positive pressure ventilatory support or of inotrope therapy. Since inotrope use was only documented until Hour 48 after surgery (end of study medication treatment), patients with inotrope use continuing until Hour 48 and with mechanical ventilation duration of ≤48 h were censored at this time point. If mechanical ventilation was continued beyond the 48-hour time point, the duration of mechanical ventilation was used in the analysis.
Time Frame: Until cessation of positive pressure ventilation and of inotrope therapy or Day 30, whichever occurred first
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Intravenous L-Citrulline | Placebo of Intravenous L-Citrulline
Number analyzed (Participants) | 11 | 11
Hours
  Re-intubation time included | 14.3 (14.06) | 44.4 (63.62)
  Re-intubation time excluded | 14.3 (14.06) | 32.0 (26.26)
Statistical Analysis 1: Comparison: Intravenous L-Citrulline vs Placebo of Intravenous L-Citrulline; Test type: Other; p = 0.0479, Wilcoxon (Mann-Whitney) — Duration including re-intubation time. Threshold for significance was p<0.05; Mean Difference (Final Values) = 30.2, 95% CI 2-sided [-10.8 to 71.1]

11. Secondary Outcome: Length of Hospitalization
Time Frame: Measured from the day of surgery until discharge from hospital or Day 30, whichever occurred first
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Intravenous L-Citrulline | Placebo of Intravenous L-Citrulline
Number analyzed (Participants) | 11 | 11
Days | 4.6 (1.21) | 8.4 (9.38)
Statistical Analysis 1: Comparison: Intravenous L-Citrulline vs Placebo of Intravenous L-Citrulline; Test type: Other; p = 0.2637, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 3.7, 95% CI 2-sided [-2.2 to 9.7]

12. Secondary Outcome: Incidence of Increased PVT (Defined as a Sustained Mean Pulmonary Artery Pressure Greater Than 20 mm Hg for at Least 2 Hours, Measured During the First 48 Hours
Description: There were insufficient data to analyze ECHO measurements in summary statistics. Additionally, most images were of very low quality and the data from ECHO evaluations were insufficient to determine whether the affected patients had pulmonary hypertension.
Time Frame: Measured in hours from the end of surgery until extubation or Day 30, whichever occurred first
Population: It was not possible to reliably determine the presence of PVT in most patients due to low quality ECHO images. Additionally, no patients were identified with sufficient ECHO measurements to detect the presence of sustained mean pulmonary artery pressure greater than 20 mm Hg for at least 2 hours.
Arm/Group | Intravenous L-Citrulline | Placebo of Intravenous L-Citrulline
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Duration of Chest Tube Drainage
Time Frame: Measured in hours from the end of surgery until removal of chest tubes or Day 30, whichever occurred first
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Intravenous L-Citrulline | Placebo of Intravenous L-Citrulline
Number analyzed (Participants) | 11 | 11
Hours | 82.7 (30.4) | 90.2 (43.7)
Statistical Analysis 1: Comparison: Intravenous L-Citrulline vs Placebo of Intravenous L-Citrulline; Test type: Other; p = 0.6431, t-test, 2 sided; Mean Difference (Final Values) = 7.5, 95% CI 2-sided [-25.9 to 41.0]

14. Secondary Outcome: Volume of Chest Tube Drainage
Time Frame: Measured in milliliters from the end of surgery until removal of chest tubes or Day 30, whichever occurred first
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Intravenous L-Citrulline | Placebo of Intravenous L-Citrulline
Number analyzed (Participants) | 11 | 11
mL | 211 (102) | 240 (257)
Statistical Analysis 1: Comparison: Intravenous L-Citrulline vs Placebo of Intravenous L-Citrulline; Test type: Other; p = 0.6408, ANOVA; Mean Difference (Final Values) = 39.5, 95% CI 2-sided [-134.2 to 213.1]

15. Secondary Outcome: Survival
Description: 28-day postoperative survival and survival to discharge
Time Frame: Measured at 28 days post surgical repair
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous L-Citrulline | Placebo of Intravenous L-Citrulline
Number analyzed (Participants) | 11 | 11
Participants | 11 | 11

16. Secondary Outcome: Number of Patients With Clinically Significant Hypotension.
Description: Age specific mean arterial blood pressure (MAP) limits compared between the citrulline and placebo groups will be used to determine significant hypotension.
  Defined as MAP below a specific age-based value (infants and age 1 year, 40; ; age 2 years, 44; age 3 years, 47; age 4 years, 50; age 5 years, 52; age 6 years, 53), that lasted greater than 30 minutes and was unresponsive to therapeutic interventions such as fluid administration (volume bolus) and increasing inotropic support.
Time Frame: Mean Arterial Blood pressure as continuously monitored postoperatively in the PCCU (Hour 0 to Hour 24) during Citrulline or Placebo infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous L-Citrulline | Placebo of Intravenous L-Citrulline
Number analyzed (Participants) | 11 | 11
Participants | 2 | 1

17. Other Pre Specified Outcome: Arginine Concentrations
Description: Citrulline is the precursor of arginine and nitric oxide. Nominal sampling times were Baseline, Post-bolus 1, Pre-bolus 2, and Hours 2, 6, 12, 24 and 48.
Time Frame: Baseline to Hour 48
Population: All randomized patients that received surgery, were treated with L-citrulline, and had at least 1 arginine concentration measurement
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Intravenous L-Citrulline | Placebo of Intravenous L-Citrulline
Number analyzed (Participants) | 11 | 11
µmol/L
  Baseline | 49.6 (15.72) | 58.7 (12.37)
  Post Bolus 1 | 72.6 (30.02) | 47.7 (7.43)
  Pre Bolus 2 | 145.1 (47.94) | 67.1 (11.66)
  Hour 6: number analyzed (Participants) | 10 | 11
  Hour 6 | 67.0 (22.66) | 47.3 (12.29)
  Hour 12: number analyzed (Participants) | 10 | 9
  Hour 12 | 61.5 (17.37) | 39.0 (12.04)
  Hour 24: number analyzed (Participants) | 10 | 9
  Hour 24 | 65.8 (18.8) | 28.1 (12.56)
  Hour 48: number analyzed (Participants) | 0 | 4
  Hour 48 |  | 34.5 (15.33)

18. Other Pre Specified Outcome: Nitric Oxide Concentrations
Description: as for outcome 17
Time Frame: Baseline to Hour 48
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Intravenous L-Citrulline | Placebo of Intravenous L-Citrulline
Number analyzed (Participants) | 11 | 11
µmol/L
  Baseline | 31.6 (13.51) | 69.5 (41.34)
  Post Bolus 1 | 25.3 (12.76) | 51.3 (38.83)
  Pre Bolus 2 | 30.7 (12.64) | 48.8 (29.16)
  Hour 6: number analyzed (Participants) | 10 | 11
  Hour 6 | 32.0 (16.97) | 59.9 (45.59)
  Hour 12: number analyzed (Participants) | 10 | 9
  Hour 12 | 26.6 (13.43) | 62.0 (42.89)
  Hour 24: number analyzed (Participants) | 10 | 9
  Hour 24 | 29.1 (12.14) | 51.1 (42.58)
  Hour 48: number analyzed (Participants) | 0 | 11
  Hour 48 |  | 42.5 (17.48)

ADVERSE EVENTS:
Time Frame: From baseline until discharge, Day 28 or early termination
Description: Obtained from signs and symptoms detected during peri- and postoperative clinical monitoring and from observations of the study personnel
Arm/Group | Intravenous L-Citrulline | Placebo of Intravenous L-Citrulline
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 8/11 | 11/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intravenous L-Citrulline (N=11) | Placebo of Intravenous L-Citrulline (N=11)
Anemia (Blood and lymphatic system disorders) | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Atrial tachycardia (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Nodal rhythm (Cardiac disorders) | 3 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 1
Pyrexia (General disorders) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Tracheitis (Infections and infestations) | 0 | 1
Blood potassium decreased (Investigations) | 1 | 2
Blood pressure systolic decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 2
Prothrombin time prolonged (Investigations) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Hemorrhage (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 4 | 3
Hypotension (Vascular disorders) | 2 | 3
Thrombosis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days